CLINICAL TRIAL: NCT06677788
Title: Efficacy and Safety of Roflumilast in Patients with Non-Alcoholic Steatohepatitis
Brief Title: Evaluating the Efficacy and Safety of Roflumilast in Patients with NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mokhtar Salem Mohamed, Doctor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35336/3/22
Record Dates: First submitted 2024-11-01; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
Keywords: NASH; Roflumilast; LSM; TNF-α; MDA; TGF-ß1
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Roflumilast; Tablets; Vitamin E

STUDY DESIGN:
Intervention Model Description: This study was a randomized controlled parallel study. Patients were recruited from out-patient clinic of Tropical medicine department, Tanta university hospital, Tanta, Egypt. The study involved 55 patients with NASH who were randomized using sealed envelope methods with assignment codes for each available allocation into vitamin E group or control group (n=24) which received vitamin E 1000 mg once daily and roflumilast group (n=31) which received roflumilast 500 μg once daily. The study duration was 3 months whereas patients were assessed at baseline and 3 months after intervention. The study was conducted following the ethical standards of Helsinki declaration in 1964 and its later amendments. The study was approved by Research Ethical committee of Tanta University (approval code:35336/3/22).participants gave their written informed consent.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Roflumilast group (n=31) (Active Comparator): Arm Description: Roflumilast group (n=31) which received roflumilast 500 μg once daily for three months. Patients were assessed at baseline and after intervention through liver stiffness measurement (LSM) using fibro-scan and through evaluation of serum levels of tumor necrosis factor -alpha (TNF-α), Malondialdehyde (MDA), transforming growth factor-beta 1 (TGF-ß1). In addition, liver enzymes, lipid panel, fasting blood glucose and fasting insulin level with subsequent calculation of homeostatic model assessment for Insulin resistance (HOMA-IR) were also assessed.
  Interventions: Drug: Roflumilast 500 Mcg Oral Tablet
- Vitamin E group or control group (n=24) (Active Comparator): vitamin E group or control group (n=24) which received vitamin E 1000 mg once daily. Patients were assessed at baseline and after intervention through liver stiffness measurement (LSM) using fibro-scan and through evaluation of serum levels of tumor necrosis factor -alpha (TNF-α), Malondialdehyde (MDA), transforming growth factor-beta 1 (TGF-ß1). In addition, liver enzymes, lipid panel, fasting blood glucose and fasting insulin level with subsequent calculation of homeostatic model assessment for Insulin resistance (HOMA-IR) were also assessed.
  Interventions: Drug: Vitamin E capsule

INTERVENTIONS:
Drug: Roflumilast 500 Mcg Oral Tablet — Patients in this group received roflumilast 500 μg once daily for three months.
  Arms: Roflumilast group (n=31)
Drug: Vitamin E capsule — vitamin E group or control group (n=24) which received vitamin E 1000 mg once daily
  Arms: Vitamin E group or control group (n=24)

SUMMARY:
Study type :clinical trial Main purpose :esnsure safety and efficacy of Roflumilast to treat patients with Non-Alcoholic Steatohepatitis Background and aim: Non-alcoholic fatty liver disease is the most prevalent chronic liver disease globally. There is no defined therapy for non-alcholic steatohepatitis (NASH), therefore this study aimed at evaluating the efficacy and safety of Roflumilast in patients with non-alcoholic NASH.

Methods: This randomized controlled parallel study involved 55 patients with NASH who were randomized into vitamin E group or control group (n=24) which received vitamin E 1000 mg once daily and roflumilast group (n=31) which received roflumilast 500 μg once daily for three months.

Patients were assessed at baseline and after intervention through liver stiffness measurement (LSM) using fibro-scan and through evaluation of serum levels of tumor necrosis factor -alpha (TNF-α), Malondialdehyde (MDA), transforming growth factor-beta 1 (TGF-ß1). In addition, liver enzymes, lipid panel, fasting blood glucose and fasting insulin level with subsequent calculation of the homeostatic model assessment for Insulin resistance (HOMA-IR) were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cytokeratine level >240 IU/L.
* Adult patient (age > 18 years old).
* Both sex.
* Overweight and obese.
* Patients with evidence of steatosis through imaging.
* Patient with mild to moderate elevation in aminotransferase activity (>2 ,but <5 times upper limit of normal ).
* Patient with Hepatic steatosis index (HSI) > 36.
* Patient with HAIR ( hypertension ,alanine aminotransferase level ,insulin resistance ) of 2 or 3.
* Fibroscan score >7Kpa and < 12.5 Kpa (F2 - F3).

Exclusion Criteria:

* Alcohol consumer and smokers
* Patients with Wilson's disease and hemochromatosis .
* Patients with viral hepatitis.
* Patients with cirrhosis .
* Patients with inflammatory diseases .
* Patients with other comorbid disease that elevate transaminases (congestive heart failure and malignancy).
* Patients on medications that interfere with lipid and carbohydrate metabolism..
* Patients on stateogenic medications.
* Pregnancy and lactating women.
* Females on oral contraceptive pills.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Change in liver stiffness measurement (LSM) measured by fibroscan score | 12 weeks following the end of treatment
  Liver Stiffness measurement (LSM) by fibro-scan. Transient elastography (Fibroscan, Echosens, Paris) was used to assess liver stiffness depending up-on the method formerly prescribed .Through a single independent operator, at least ten valid measurements were obtained for each patient. Results were included in the final analysis only if the following three criteria were met: at least ten valid measurements, success rate >60% and the interquartile range (IQR)-to-liver stiffness ratio was ≤0.30. The median values of the validated measurements for each patient were representative to the liver stiffness and expressed in units of kilopascals (kPa)

SECONDARY OUTCOMES:
The change in liver panel parameters | 3 months after treatment
  Blood sample collection and biochemical measurement of Approximately 10 ml of venous blood was taken from each patient after overnight fasting by sterile venipuncture, without frothing and after minimal venous stasis using disposable syringes. Blood samples were delivered in a vacutainer serum separator tubes. Immediate centrifugation at 3000 rpm was performed and then the serum was separated and divided into two portions. The first portion was used for determination of fasting blood glucose (glucose oxidase method), liver enzymes aspartate transaminase "AST", alanine transaminase "ALT" and gamma-glutamyl transaminase "GGT" (spectrophotometerially) and lipid panel (enzymatic colorimeteric method).
Improvement in HOMA IR | 12 weeks following the end of treatment
  HOMA-IR is calculated as [Fasting Insulin (μg/ml)]*[Fasting Glucose (mmol/l)]/22.5,HOMA-IR values between 0.5 and 1.4 are considered normal, ≥1.9 are indicative of early IR, and ≥2.9 indicate IR

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Mohamed Mostafa, Professor of clinical pharmacy, Study Chair — Faculty of Pharmacy , Tanta University, Tanta, Egypt
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in non alcoholic steatohepatitis. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact Mokhtaarsalem@gmail.com